CLINICAL TRIAL: NCT05775679
Title: Test-Retest Reliability, Responsiveness and Interpretability of CLEFT-Q
Acronym: CLEFT-QSwePsyc
Status: Recruiting | Type: Observational
Sponsor: Department of Plastic and Reconstructive Surgery (Network)
Collaborators: Karolinska University Hospital (Other); Linköping Univeristy Hospital (Unknown); Umeå University Hospital (Unknown); Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-06993-01
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Cleft Lip and Palate
Keywords: CLEFT-Q; Psychometrics; Test-retest reliability; Interpretability; Responsiveness
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Test-retest reliability: 50 patients answer CLEFT-Q twice with 1-2 weeks in between.
- Secondary Nose Surgery: 50 patients answer CLEFT-Q before and 6 months after secondary nose surgery.
- Secondary Lip Surgery: 50 patients answer CLEFT-Q before and 6 months after secondary lip surgery.
- Jaw Surgery: 50 patients answer CLEFT-Q before and 1 year after jaw surgery.
- Secondary Speech Improving Surgery: 50 patients answer CLEFT-Q before and 1 year after secondary speech improving surgery.
- Health care professionals: 20 health care professionals will be interviewed about their experiences on working with CLEFT-Q.

SUMMARY:
The goal of this observational study is to test the questionnaire CLEFT-Q in a population of patients with cleft lip and/or palate. The main questions it aims to answer are:

1. Are CLEFT-Q scores reliable over time?
2. Can CLEFT-Q detect change following surgical treatment intervention?
3. What is the norm for CLEFT-Q within a control population who do not have cleft lip and/or palate?
4. What is the Minimal Clinically Important Change of CLEFT-Q in different subpopulations of cleft lip and/or palate?
5. Do changes in CLEFT-Q scores correlate with changes in objective outcomes following a surgical intervention?
6. What are the main expectations that patients express before a surgical intervention?
7. How do patients perceive that the results after surgical interventions meet their expectations?
8. Do patients express concepts of importance postoperatively that are not examined by CLEFT-Q?
9. How do healthcare professionals perceive that the use of CLEFT-Q affects clinical decisions and processes?

Participants will

1. Fill out the questionnaire CLEFT-Q twice with a two-week space.
2. Before and 1 year after an operation.
3. Be interviewed about their experiences related to an operation or using CLEFT-Q.

Researchers will compare results from the cleft lip and palate population to see if there is a difference between them and a population without cleft lip and palate.

ELIGIBILITY:
Inclusion Criteria:

* Cleft lip and/or palate
* Planned secondary surgery of the nose, lips, jaw or to improve speech
* Can speak and read Swedish

Exclusion Criteria:

* Multiple surgeries at once

Ages: 8 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: - Patients with cleft lip and/or palate who have been operated as infants and opt for secondary surgery to improve appearance, occlusion or speech.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
CLEFT-Q change scores | At enrollment and after 1-2 weeks, or after 6 months, or after 1 year.
  CLEFT-Q is a questionnaire on health related quality of life specific to patients with cleft lip and palate

SECONDARY OUTCOMES:
Photograph | Before surgery and after 6 months or 1 year.
  Photographs from before and after surgery
Speech | Before surgery and after 1 year.
  Recording of speech

CONTACTS AND LOCATIONS:
Overall Officials: Mia Stiernman, MD PhD, Principal Investigator — Mia Stiernman
Locations (1):
- Skania University Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided